CLINICAL TRIAL: NCT06163690
Title: Digital Symptom Tracking and Wellness in Long COVID Patients Using Endourage Targeted Wellness Formula C™ Sublingual Drops
Brief Title: Symptom Tracking in Long COVID Patients Using Formula C™ Sublingual Drops
Status: Completed | Type: Observational
Sponsor: Endourage, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Endo2023
Record Dates: First submitted 2023-12-07; First posted 2023-12-11 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-10

CONDITIONS: Long COVID; Long Covid19; Post-Acute COVID-19; Post-Acute COVID-19 Syndrome; Long Haul COVID; Long-Haul COVID-19
Keywords: Hemp; Terpenes; Cannabinoids; Entourage effect
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Endourage Targeted Wellness Formula C™, a full hemp flower extract — A hemp-derived formulation designed as a daily use adjunctive therapy to help improve Long COVID symptoms. Endourage Targeted Wellness Formula C™ are used as sublingual drops held under the tongue for 60 to 90 seconds.

SUMMARY:
This is a digital symptom tracking study of Formula C™, a full cannabis flower formulation, rich in cannabinoids and terpenes, that has been shown to improve symptoms in people with Long COVID. Participants 21 and older will take Formula C™ for 90 days. During that time, participants will answer weekly surveys to track symptoms and wellbeing.

DETAILED DESCRIPTION:
Long COVID is a global health crisis with no current treatments. There's a growing interest within the medical community to explore the potential benefits of full hemp flower extracts in treating and alleviating Long COVID symptoms. Full hemp flower extracts are a remarkable advancement in the field of natural wellness and healing. Full hemp flower extracts harness the full spectrum of beneficial compounds present in the hemp plant, including not just cannabidiol (CBD), but a host of other cannabinoids, terpenes, and flavonoids. This process, known as 'whole plant' or 'full spectrum' extraction, produces a more potent and therapeutic product, as the various compounds work synergistically in what is referred to as the 'entourage effect'. These extracts have been associated with a broad range of potential health benefits, such as pain relief, reduction of inflammation, anxiety management, and sleep improvement. A recently published single-blind, randomized, placebo controlled trial demonstrated that Long COVID patients benefitted from sublingual use of Formula C without any safety events. This remote, observational study of Endourage Targeted Wellness Formula C™ sublingual drops will seek to empower participants to track symptoms and wellbeing while taking Formula C to determine if Long COVID symptoms are attenuated and time to healing is shortened.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 21 years of age.
2. Willing and able to read, understand, and sign the informed consent.
3. Willing to comply with all study procedures.
4. Must have device to access the internet to complete surveys online.
5. A diagnosis of Long COVID from a health care provider.

Exclusion Criteria:

1. Non-English speaking, as the surveys are developed in the English language.
2. Known allergies to hemp seeds or hemp-derived products, medical cannabis, coconut oil.
3. Pregnancy, or planning to become pregnant in the next 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People located in the U.S. that have been diagnosed with Long COVID and are being treated by a physician for Long COVID symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Symptom and wellbeing change over 3 months | 90 days
  This study will use the PROMIS-29+2 Profile v2.1 (PROPr) is used to calculate a change in Long COVID related symptoms including fatigue, sleep, pain, mood and physical function.

SECONDARY OUTCOMES:
Patient Global Impression of Change | 90 days
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Steward, MD, Principal Investigator — Endourage, LLC
Locations (1):
- Endourage, LLC, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young TP, Erickson JS, Hattan SL, Guzy S, Hershkowitz F, Steward MD. A Single-Blind, Randomized, Placebo Controlled Study to Evaluate the Benefits and Safety of Endourage Targeted Wellness Formula C Sublingual +Drops in People with Post-Acute Coronavirus Disease 2019 Syndrome. Cannabis Cannabinoid Res. 2024 Feb;9(1):282-292. doi: 10.1089/can.2022.0135. Epub 2022 Oct 14. PMID 36252151